CLINICAL TRIAL: NCT07036718
Title: A Prospective, Non-interventional Study to Evaluate the Efficacy and Safety of Iptacopan in Adults With Paroxysmal Nocturnal Hemoglobinuria (PNH) in Routine Clinical Practice in the Russian Federation
Brief Title: NIS PDC the Efficacy and Safety of Iptacopan in Adults in Routine Clinical Practice
Acronym: PRIORITY- PNH
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLNP023C1RU03
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH; Paroxysmal nocturnal hemoglobinuria; Iptacopan
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- iptacopan: Adults with PNH who started the iptacopan therapy

SUMMARY:
This is a prospective, non-interventional, multicenter study to evaluate the efficacy and safety of iptacopan in patients with PNH in real-world settings in Russia.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the start of iptacopan therapy.
2. The patient is undergoing treatment with iptacopan.
3. The treating physician decided to prescribe iptacopan based on the Summary of Product Characteristics during routine clinical practice, regardless of study participation.
4. Provision of written informed consent.

Exclusion Criteria:

1. Any situations where iptacopan is contraindicated in accordance with the Summary of Product Characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment of female and male patients with PNH
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with an increase in Hb level ≥ 20 g/l | 6 months
  Number of patients who achieved an increase in Hb level ≥ 20 g/l over 6 months after iptacopan treatment initiation and were Red Blood Cells (RBC) transfusion independent.

SECONDARY OUTCOMES:
Number of patients with an increase in Hb level ≥ 120 g/L | 12 months
  Number of patients who achieved an increase in Hb level ≥ 120 g/L at 12 months after initiation of iptacopan treatment and were RBC transfusion independent
Number of patients with an increase in Hb level ≥ 20 g/L | 12 months
  Number of patients who achieved an increase in Hb level ≥ 20 g/L at 12 months after initiation of iptacopan treatment and was RBC transfusion independent
Change from baseline in reticulocyte count (10⁹/L) | 12 months
  Change from baseline in reticulocyte count (10⁹/L) over 12 months after initiation of iptacopan treatment
Change from baseline in LDH levels (U/L) | 12 months
  Change from baseline in LDH levels (U/L) over 12 months after initiation of iptacopan treatment
Number of patients with an absence of administration of packed-RBC transfusions | 12 months
  Number of patients with an absence of administration of packed-RBC transfusions at 12 months after initiation of iptacopan treatment
Change from baseline in the Hb level (g/L) | Baseline, month 3, month 6 and month 12
  Change from baseline in the Hb level (g/L) at 3, 6 and 12 months after initiation of iptacopan treatment
Number of breakthrough hemolysis (BTH) | 12 months
  Number of breakthrough hemolysis (BTH) cases 12 months following the initiation of iptacopan therapy
Percentage of patients by BMI | 12 months
  Percentage of patients by Body mass index (BMI) (<25, 25.1-29.9, >30)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Russia (7):
  - Novartis Investigative Site, Syktyvkar, Komi
  - Novartis Investigative Site, Grozny
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Murmansk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yuzhno-Sakhalinsk

IPD SHARING:
Plan to Share IPD: No